CLINICAL TRIAL: NCT07208773
Title: A Multi-center, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Preliminary Efficacy of YL201 in Combination With Ivonescimab in Patients With Advanced Solid Tumors
Brief Title: A Study of YL201 and Ivonescimab (AK112) in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Akesobio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-104-02
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors; Non Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: Advanced solid tumors; PD1/VEGF Bispecific; Antibody drug conjugate; Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1： Safety run-in (Experimental): Multiple dose levels of YL201 will be explored in combination with Ivonescimab administered intravenously (IV) at a fixed dose.Participants receive YL201 and Ivonescimab (AK112) on Day 1 of each 3-week cycle, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: YL201; Drug: Ivonescimab
- Phase 2： Dose expansion (Experimental): YL201 will be administered at the selected RDE in combination with Ivonescimab administered IV at a fixed dose. Participants receive YL201+ Ivonescimab (AK112) on Day 1 of each 3-week cycle, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: YL201; Drug: Ivonescimab

INTERVENTIONS:
Drug: YL201 — YL201 will be administered as IV infusion
Drug: Ivonescimab — Ivonescimab will be administered as IV infusion.

SUMMARY:
This study was designed to evaluate the efficacy and safety of YL201 in combination with Ivonescimab (AK112) in subjects with solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Inclusion criteria for the study population： Phase 1: Advanced Solid tumors. Phase 2: Extensive-stage SCLC, Non-AGA NSCLC, EGFR mutation NSCLC.
3. ECOG PS score is 0 or 1.
4. Within 7 days before the first dose, the functions of body organs and bone marrow meet the requirements.

Exclusion Criteria:

1. Suitable for local curative treatment.
2. Have received previous treatment with drugs targeting B7-H3 (including antibodies, ADCs, CAR-T, and other drugs).
3. Have received previous treatment with topoisomerase I inhibitors or ADCs containing topoisomerase I inhibitors.
4. Have experienced grade ≥ 3 irAEs during previous treatment with anti-programmed death receptor (ligand) [anti-PD-(L)1] or other immune checkpoint inhibitors.
5. History of bleeding tendency or coagulation disorders and/or clinically significant bleeding symptoms or risks within 4 weeks before randomization.
6. Imaging studies during the screening period show that the patient has the Imaging-confirmed tumor invasion of major blood vessels.
7. Active autoimmune disease requiring systemic treatment.
8. Brain metastases or spinal cord compression.
9. Patients with uncontrolled or clinically significant cardiovascular diseases.
10. Clinically significant concurrent pulmonary diseases.
11. Known to have active pulmonary tuberculosis. Other protocol-defined inclusion/ exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Approximately within 36 months
  AEs are assessed based on NCI CTCAE v5.0.
Maximum tolerate dose（MTD) | Approximately within 36 months
Recommended Dose for Expansion | Approximately within 36 months
Objective Response Rate (ORR) | Approximately within 36 months
  ORR defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) | Approximately within 36 months
maximum concentration (Cmax) | Approximately within 36 months
minimum concentration at trough (Ctrough) | Approximately within 36 months
Volume of distribution (Vd) | Approximately within 36 months
plasma clearance (CL) | Approximately within 36 months
half-life (t1/2) | Approximately within 36 months
Time to peak drug concentration (Tmax) | Approximately within 36 months
Investigator-assessed progression-free survival (PFS) | Approximately within 36 months
  PFS defined as the time interval from the first study drug administration to the first documented PD or death due to any cause, whichever occurs first
Investigator-assessed overall survival (OS) | Approximately within 36 months
  OS defined as the time interval from the first study drug administration to death due to any cause.
Investigator-assessed disease control rate (DCR) | Approximately within 36 months
  DCR defined as the proportion of subjects with a BOR of CR, PR, or stable disease (SD).
Investigator-assessed time to response (TTR) | Approximately within 36 months
  TTR defined as the time interval from the first study drug administration to the first documentation of response (CR or PR).
Investigator-assessed the depth of response (DpR) per RECIST v1.1 | Approximately within 36 months
  The percentage change in target lesion size
number of subjects who are Anti-Drug Antibody (ADA)-positive at any time | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China